CLINICAL TRIAL: NCT03408847
Title: Supplementation of Extra Virgin Olive Oil Monocultivar Coratina in Patients With Active Ulcerative Colitis
Brief Title: Monocultivar Coratina Extra Virgin Olive Oil in UC Patients
Acronym: EVORCU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Collaborators: Fondazione Schena (Other)
Responsible Party: Principal Investigator, Angelo Andriulli, Medical Doctor, Casa Sollievo della Sofferenza IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EVO-RCU-2017
Record Dates: First submitted 2017-11-24; First posted 2018-01-24 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Ulcerative Colitis Chronic Mild
Keywords: Ulcerative colitis; UC; Extra virgin olive oil; Polyphenols
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Beclomethasone

STUDY DESIGN:
Intervention Model Description: Pilot study
Who Masked: Participant, Investigator
Masking Description: Patients will receive a bottle with experiental oil or placebo, consisting of commercial refined olive oil. No diffencences between the two bottles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MC-EVOO in addition to steroid therapy (Active Comparator): Oral beclomethasone dipropionate at dose of 10 mg / day for the first 4 weeks, 5 mg / day for the second 4 weeks plus MC- EVOO for 12 weeks at a dose of 2 tablespoons per day (1 before lunch and 1 before dinner). Each spoon will contain 10 grams of oil containing 5 mg of biophenols.
  Interventions: Combination Product: Beclomethasone dipropionate in addition to MC-EVOO
- Refined olive oil and steroid therapy (Placebo Comparator): Oral beclomethasone dipropionate (10 mg / day for the first 4 weeks, 5 mg / day for the second 4 weeks) plus placebo consisting of refined olive oil with low biophenols.
  Interventions: Combination Product: Beclomethasone dipropionate in addition to refined oil

INTERVENTIONS:
Combination Product: Beclomethasone dipropionate in addition to MC-EVOO — Oral beclomethasone dipropionate at dose of 10 mg / day for the first 4 weeks, 5 mg / day for the second 4 weeks plus MC- EVOO for 12 weeks at a dose of 2 tablespoons per day (1 before lunch and 1 before dinner). Each spoon will contain 10 grams of oil containing 5 mg of biophenols.
  Arms: MC-EVOO in addition to steroid therapy
Combination Product: Beclomethasone dipropionate in addition to refined oil — Oral beclomethasone dipropionate (10 mg / day for the first 4 weeks, 5 mg / day for the second 4 weeks) plus placebo consisting of refined olive oil with low biophenols.
  Arms: Refined olive oil and steroid therapy

SUMMARY:
Epidemiological studies suggest that daily intake of fruits and vegetables high in polyphenols or the addition of olive oil containing many polyphenols is associated with a reduced risk of chronic diseases including cardiovascular, metabolic, neurodegenerative, and inflammatory bowel conditions.

In vivo experiments demonstrated that the administration of a diet associated with daily intake of extra virgin olive oil (EVOO) reduces histological lesions and symptomatology in rats with a dextran sulfate sodium (DDS) induced colitis. A diet supplemented with hydroxytyrosol (a component of olive oil) showed a reduction of the inflammatory process at the inflamed colon of the rats.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease of unknown etiology, which usually occurs in young adults (II-IV decade of life).

Epidemiological data have shown a north-south gradient of both incidence and prevalence of UC in European countries, with a higher prevalence in northern European countries than in the Mediterranean area. However, recent data show a reduction in these differences in the last two decades. The reasons of this reduction are unknown, but it is possible that these differences are related to a change in dietary habits in southern European countries where a diet rich in fresh fruits and vegetables (the so-called "Mediterranean diet") is gradually being replaced by a typical diet of the industrialized countries of northern Europe, characterized by high consumption of frozen or pre-packaged foods of the food industry.

These changes in the diet regime have also replaced the type of oil contained in foods, ranging from olive oil (typical of the Mediterranean diet) to fats of animal origin or vegetable oils not coming from the olives.

Olive oil is universally recognized as the symbol of the Mediterranean diet and its beneficial properties have been extensively studied.

In particular, there are scientific evidence showing an effect of virgin olive oil on the lipid metabolism, on chronic inflammation, on blood pressure, and the regulation and detoxification of free radicals.

In particular, beneficial effects would in part be related to polyphenols, potent natural antioxidants contained in olive oil.

Monocultivar Coratina extra virgin olive oil (MC-EVOO) is an Apulian olive oil that, while possessing an extraordinary health effect superior to other cultivars, is not very used because of its distinctive characteristics of bitter and spicy. The bitter and the spicy of the extra virgin olive oil obtained from Coratina monocultivar are not defects in the oil but are the expression of a very high concentration of polyphenols (up to 800-1000 mg / kg of oil) compared to other varieties which, as well as providing extraordinary health benefits to the consumer, extend the expiration date of the oil itself, preserving it from oxidative action.

The MC-EVOO is a typical of the Apulia Region and it is characterized by:

1. high content of polyphenols
2. natural 100% product, with no residues of chemical solvents and other toxic and harmful contaminants.

No studies have been published so far that have demonstrated a potential toxic effects of polyphenols. Instead, EVOO-C supplementation could potentially have positive effects on lipid metabolism and body weight.

Epidemiological studies suggest that daily intake of fruits and vegetables high in polyphenols or the addition of olive oil containing many polyphenols is associated with a reduced risk of chronic diseases including cardiovascular, inflammatory, metabolic, neurodegenerative, and some neoplasms.

Also the results of in vitro study showed these properties but these results have to be carefully evaluated because in vivo the polyphenols, after being absorbed into the intestine and conjugated in the liver, arrive in the blood in methylated, sulphated and glycogenated form.

These molecules are completely different from the structural point of view of native molecules. Moreover, their presence is in the concentration of nano or micro molecules. These molecules have different biological properties from native ones and are distributed differently in different tissues and cells.

In addition, in the in-vitro studies native polyphenol molecules have been used at high concentrations, or above physiological (over 100 micromoles).

This is the first reason why a clinical trial case study was planned. Polyphenols also modulate cell membranes, enzymes, transcription factors and receptors. This is the second reason why nutrigenomics will be studied during the course of the clinical trial to evaluate the effects of polyphenols on the molecular and cellular mechanisms of the inflammatory processes that are present in the ulcerative colitis.

In vivo experiments demonstrated that the administration of a diet associated with daily intake of EVOO reduces histological lesions and symptomatology in rats with a DDS induced colitis. A diet supplemented with hydroxytyrosol (a component of olive oil) showed a reduction of the inflammatory process at the inflamed colon of the rats.

These data show that EVOO supplementation in a diet can improve the course of the disease.

Experimental studies in humans are limited. The first study published over 25 years ago concluded that administering a supplement of fish oil to the diet produced a modest reduction in corticosteroid in the active phases of the disease, but not a benefit in maintenance therapy over olive oil. This work presents important limitations:

1. the content of polyphenols in the oils used is unknown
2. the remission time between the two oils was not statistically significant
3. there are no data on inflammation of the colon before and after treatment Recently, an in vitro study performed on intestinal mucosa obtained from 14 active UC patients showed that samples treated with oleuropein had a reduced expression of two inflammatory factors, COX-2 and IL-17, suggesting that olive oil containing oleuropein can improve inflammatory status.

The aim of the study is to evaluate whether MC- EVOO supplementation in moderate to severe UC patients needing a steroid cycle may increase the clinical response rate to medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active UC (diagnosed for at least 3 months) aged 18 to 70 years
* Patients with mild to moderate disease (calculated by Mayo score).
* Patients can provide their informed consent to participate in the study

Exclusion Criteria:

* Patients with Crohn's disease
* Patients with complicated disease, who are candidates for urgent surgery
* Patients with colostomy
* Patients with contraindications to steroid therapy (diabetes mellitus, severe osteoporosis, vertebral fractures, previous intolerance to steroid therapy)
* Patients with unstable or inappropriately controlled cardiovascular, pulmonary, hepatic, renal or hematologic diseases
* Patients who are not compliant
* Patients abusing alcohol or drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the short-term clinical response | 12 weeks
  Evaluation of the short-term clinical response rate in the 2 treatment groups

SECONDARY OUTCOMES:
Evaluation of the clinical remission | 12 weeks
  Evaluation of the clinical remission rate in the short term in the 2 treatment groups
Evaluation of the endoscopic remission | 12 weeks
  Evaluation of the endoscopic remission rate after 3 months in the 2 treatment groups
Evaluation of markers of inflammation | 12 weeks
  Evaluation of the rate of patients with normalization of markers of inflammation in the short and medium term in the 2 treatment groups
Evaluation of adverse events | 12 weeks
  Evaluation of the rate of adverse events in the 2 treatment groups

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danese S, Fiocchi C. Ulcerative colitis. N Engl J Med. 2011 Nov 3;365(18):1713-25. doi: 10.1056/NEJMra1102942. No abstract available. PMID 22047562
- [Background] Ng SC, Bernstein CN, Vatn MH, Lakatos PL, Loftus EV Jr, Tysk C, O'Morain C, Moum B, Colombel JF; Epidemiology and Natural History Task Force of the International Organization of Inflammatory Bowel Disease (IOIBD). Geographical variability and environmental risk factors in inflammatory bowel disease. Gut. 2013 Apr;62(4):630-49. doi: 10.1136/gutjnl-2012-303661. Epub 2013 Jan 18. PMID 23335431
- [Background] Koloski NA, Bret L, Radford-Smith G. Hygiene hypothesis in inflammatory bowel disease: a critical review of the literature. World J Gastroenterol. 2008 Jan 14;14(2):165-73. doi: 10.3748/wjg.14.165. PMID 18186549
- [Background] Sanchez-Fidalgo S, Sanchez de Ibarguen L, Cardeno A, Alarcon de la Lastra C. Influence of extra virgin olive oil diet enriched with hydroxytyrosol in a chronic DSS colitis model. Eur J Nutr. 2012 Jun;51(4):497-506. doi: 10.1007/s00394-011-0235-y. Epub 2011 Aug 27. PMID 21874330
- [Background] Takashima T, Sakata Y, Iwakiri R, Shiraishi R, Oda Y, Inoue N, Nakayama A, Toda S, Fujimoto K. Feeding with olive oil attenuates inflammation in dextran sulfate sodium-induced colitis in rat. J Nutr Biochem. 2014 Feb;25(2):186-92. doi: 10.1016/j.jnutbio.2013.10.005. Epub 2013 Nov 8. PMID 24445043
- [Background] Reddy KVK, Naidu KA. Oleic acid, hydroxytyrosol and n-3 fatty acids collectively modulate colitis through reduction of oxidative stress and IL-8 synthesis; in vitro and in vivo studies. Int Immunopharmacol. 2016 Jun;35:29-42. doi: 10.1016/j.intimp.2016.03.019. Epub 2016 Mar 24. PMID 27016717
- [Background] Hawthorne AB, Daneshmend TK, Hawkey CJ, Belluzzi A, Everitt SJ, Holmes GK, Malkinson C, Shaheen MZ, Willars JE. Treatment of ulcerative colitis with fish oil supplementation: a prospective 12 month randomised controlled trial. Gut. 1992 Jul;33(7):922-8. doi: 10.1136/gut.33.7.922. PMID 1353742
- [Background] Larussa T, Oliverio M, Suraci E, Greco M, Placida R, Gervasi S, Marasco R, Imeneo M, Paolino D, Tucci L, Gulletta E, Fresta M, Procopio A, Luzza F. Oleuropein Decreases Cyclooxygenase-2 and Interleukin-17 Expression and Attenuates Inflammatory Damage in Colonic Samples from Ulcerative Colitis Patients. Nutrients. 2017 Apr 15;9(4):391. doi: 10.3390/nu9040391. PMID 28420140